CLINICAL TRIAL: NCT03526796
Title: Hyperbaric Oxygen Therapy for Antibiotic Refractory Pouchitis: a Phase 2A Clinical Trial
Brief Title: Hyperbaric Oxygen Therapy for Antibiotic Refractory Pouchitis
Acronym: HBOT-pouch
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jinling Hospital, China (Other)
Responsible Party: Principal Investigator, Jianfeng Gong, Associate Professor, Jinling Hospital, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HBOT-pouchitis
Record Dates: First submitted 2018-04-14; First posted 2018-05-16 (Actual); Last update posted 2018-05-16 (Actual); Status verified 2018-05

CONDITIONS: Pouchitis; Hyperbaric Oxygen Therapy
Keywords: Pouchitis; Hyperbaric oxygen therapy
MeSH Terms: conditions — Pouchitis | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hyperbaric oxygen therapy (Experimental): Patients who recieve hyperbaric oxygen therapy will be maintained at 2.4 ATA with 100% oxygen for 90 min and then decompressed back to 1 ATA. The treatment duration is 4 weeks and extends to 6 weeks if necessary.
  Interventions: Procedure: Hyperbaric oxygen therapy

INTERVENTIONS:
Procedure: Hyperbaric oxygen therapy — Patients were maintained at 2.4 ATA with 100% oxygen for 90 min and then decompressed back to 1 ATA. The treatment duration is 4 weeks and extends to 6 weeks if necessary.

SUMMARY:
The aim of current study is to evaluate the effect of hyperbaric oxygen therapy for the treatment of chronic antibiotic-refractory pouchitis.

DETAILED DESCRIPTION:
Pouch ischemia plays an important role in the pathogenesis of pouchitis after IPAA surgery for ulcerative colitis. Obese Male patients are at high risk for pouchitis because of mesenteric tension. Excessive weight gain is associated with an increased risk for pouch failure in patients with restorative proctocolectomy. Also, patients with an 'S' pouch hardly ever develop chronic pouchitis, owing to the additional length of bowel loop along with mesentery when attached to the anal transitional zone. The treatment of chronic antibiotic-refractory pouchitis(CARP) is difficult.

Hyperbaric oxygen therapy(HBOT) have been proven effecitve in the treatment of inflammatory bowel diseases(IBD). Meta-analysis revealed that the overall response rate was 86% (85% CD, 88% UC), and of the endoscopic response rate to HBOT is 100%. The possible mechanism might be due to the prmoted wound healing by increasing oxygen delivery to hypooxic tissues and changes in inflammatory and immunological mediators.

Therefore, the aim of current study is to examine the therapeutic effect of HBOT for chronic antibiotic-refractory pouchitis(CARP).

ELIGIBILITY:
Inclusion Criteria:

* IPAA performed for ulcerative colitis;
* Pouchitis Disease Activity Index (PDAI) scores ≥7;
* Antibiotic refractory pouchitis(CARP), defined as patients who do not respond to conventional 2-week, single-agent antibiotic therapy including metronidazole,ornidazole,tinidazole, or ciprofloxacin
* 18-75years
* Informed consent given
* Able and willing to comply with all trial procedures
* Including prepouch ileitis

Exclusion Criteria:

* Crohn's disease of the pouch
* Pouchitis after IPAA for FAP
* Isolated cuffitis
* with cocomttant Primary sclerosing cholangitis (PSC)
* Pouch strictures
* Abscess/Sinuses
* Perianal disease
* Active malignancy
* Uncontrolled systemic diseases
* History of noninfammatory disease of the pouch
* Decreased pouch compliance
* Irritable pouch syndrome
* Afferent or efferent limb obstruction
* Needing oral or topical steroid or 5-ASA
* Major physical or psychiatric illness within the last 6m
* Active use of cholestyramine, NSAIDs or aspirin
* Pregnant, breast feeding
* Clinically significant co-morbidities causing untolerant or unsuitable for hyperbaric oxygen therapy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-06-01 (Estimated); Primary Completion 2020-05 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Remission rate | up to 4 weeks
  Defined by a pouchitis disease activity index (PDAI) score of < 7 points

SECONDARY OUTCOMES:
Response rate | up to 4 weeks
  Defined as a ≥ 3-point reduction in the 18-point PDAI scoring system
Symptomatic improvement rate | up to 4 weeks
  Reduction of PDAI clinical subscore >2 points.
Endoscopic improvement rate | up to 4 weeks
  Reduction of PDAI endoscopic subscore >2 points.
Fecal calprotectin level | up to 4 weeks
  Fecal caprotectin level before and after treatment
Plasma C-reactive protein level | up to 4 weeks
  Plasma caprotectin level before and after treatment
Plasma Interleukin-6 level | up to 4 weeks
  Plasma Interleukin-6 level before and after treatment
Fecal microbiome | up to 4 weeks
  Fecal microbiome analysis using 16S RNA technique before and after treatment
Adverse events | up to 4 weeks
  Any adverse event deemed as possibly, probably, or definitely related to investigational treatment during 2-3 weeks of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Jianfeng Gong, MD, Principal Investigator — Jinling Hospital, China
Locations (1):
- Department of Generay Surgery, Jinling hosptal, Medical School of Nanjing University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided